CLINICAL TRIAL: NCT06187363
Title: Tubularized Incised Plate (TIP) Procedure Versus Other Procedures in the Repair of Disrupted Hypospadias
Brief Title: Redo Repair in Disrupted Hypospadias
Status: Completed | Type: Observational
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Ahmed Elrouby, Associate Professor of pediatric Surgery, Egyptian Biomedical Research Network
Other Study IDs: 0306287
Record Dates: First submitted 2023-09-22; First posted 2024-01-02 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hypospadias
Keywords: Hypospadias; Redo repair; Disruption
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients managed by tubularized incised plate procedure: Patients with redo hypospadias repair using tubularized incised plate procedure
  Interventions: Procedure: Tubularized incised plate procedure
- Patients treated by procedures other than tubularized incised plate procedure: Patients with redo hypospadias repair using other procedures
  Interventions: Procedure: Other procedures

INTERVENTIONS:
Procedure: Tubularized incised plate procedure — Tubularized incised plate urethroplasty procedure
  Groups: Patients managed by tubularized incised plate procedure
Procedure: Other procedures — Other procedures than tubularized incised plate urethroplasty procedure
  Groups: Patients treated by procedures other than tubularized incised plate procedure

SUMMARY:
Redo hypospadias repair is a challenging situation and its success depends on many factors. Several procedures could be used in such situations with variable outcomes. The investigator in this study aimed at comparing the results of these procedures

DETAILED DESCRIPTION:
Purpose: Our study compared the outcome of the tubularized incised plate urethroplasty procedure and other procedures in the case of redo hypospadias repair. Methods: The participants were categorized into those who were treated by the tubularized incised plate procedure (Group A) and those who were treated by other procedures (Group B) and the collected data were compared between the two groups. The patients were examined regularly during the postoperative period for urethral-cutaneous fistula, meatal stenosis, penile curvature, penile skin coverage, and re-disruption.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with disrupted hypospadias repair

Exclusion Criteria:

* Fresh cases of hypospadias

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fifty patients were included in our study; all of them have disrupted repair of hypospadias. Half of those patients were treated by TIP procedure and the other half were treated by other procedures
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The number of participants who developed post-operative meatal stricture | at 1 month, 3 months, 6 months, and at the end of the 1st year
  assessment of the position of neo-meatus in glans together with its diameter as well as the presence of stenosis as judged by urethral calibration
The rate of development of recurrent post-operative chordae | at 1 month, 3 months, 6 months, and at the end of the 1st year
  The recurrence of ventral penile chordae as discovered by recurrent ventral penile curvature
The incidence of development of postoperative penile skin scarring | at 1 month, 3 months, 6 months, and at the end of the 1st year
  Assessment of penile skin coverage as judged by the development of recurrent curvature, torsion and/or disfigurement
The incidence of the development of failed repair as discovered by the position of the neo-meatus | at 1 month, 3 months, 6 months, and at the end of the 1st year
  Re-disruption the reposition of the neo-meatus to the previous site
The incidence of the development of post-operative urethral-cutaneous fistula | at 1 month, 3 months, 6 months, and at the end of the 1st year
  The development of post-operative urethral-cutaneous fistula as judged by the development of a second urethral openning proximal to the neo-meatus

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elrouby, MD, Principal Investigator — Pediatric Surgery department
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No